CLINICAL TRIAL: NCT06394895
Title: Donor Neutrophil Subsets to Predict the Risk of Acute Graft-versus-Host Disease Following Allogeneic Hematopoietic Stem Cell Transplantation
Brief Title: Donor Neutrophil Subsets to Predict the Risk of aGVHD
Status: Active, not recruiting | Type: Observational
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: NFEC-2023-500
Record Dates: First submitted 2023-12-20; First posted 2024-05-01 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Acute Graft-versus-Host Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 100 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Subject-recipient (high incidence /low incidence group)
- Subject-donor

SUMMARY:
This is a prospective study to explore the association between donor neutrophil subsets and acute graft-vs.-host disease outcomes. Approximately 260 subjects (including 130 donors and 130 corresponding recipients) will be recruited.

DETAILED DESCRIPTION:
This study was a single-center, observational, prospective cohort study. The study lasted for 3 months, from 2023.12 to 2024.3, the clinical enrollment was completed, and from 2024.3 to 2024.6, the follow-up was completed. It is planned to enroll 260 subjects, divided into 130 donors and 130 patients.

No randomization or any protocol-driven treatment will be performed or provided to subjects during the course of the study. Treatment decisions and selection of treatment options are left to the discretion of the treating physician, if clinically appropriate.

All recipients will be followed for aGVHD evaluation, relapse, cGVHD, leukemia relapse, disease-free survival (DFS), non-relapse mortality (NRM). aGVHD and cGVHD were graded according to published guidelines. All recipients will be monitored every month until the study is completed.

ELIGIBILITY:
Inclusion Criteria:

Donors

1. Voluntarily sign the informed consent form;
2. Age 16-65 years old
3. Donors whose HLA-matched or HLA-mismatched to the corresponding recipients

Recipients

1. Voluntarily sign the informed consent form
2. Age 16-65 years old
3. Willing to undergo HLA-matched or HLA-mismatched allo-HSCT

Exclusion Criteria:

Donors

1. Have a history of other tumors
2. With poor compliance or mental disorders
3. Infected with HIV and HCV
4. With uncontrolled HBV infection
5. With other autoimmune diseases
6. Those who are judged by the researcher to be unsuitable to participate in this study

Recipients

1. Have a history of other tumors
2. With poor compliance or mental disorders
3. Infected with HIV and HCV
4. With uncontrolled HBV infection
5. With other autoimmune diseases
6. Those who are judged by the researcher to be unsuitable to participate in this study

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients following allogeneic hematopoietic stem cell transplantation and the corresponding donors
Sampling Method: Non-Probability Sample
Enrollment: 260 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-02-29 (Actual); Study Completion 2024-06-10 (Estimated)

PRIMARY OUTCOMES:
Association between donor neutrophil subsets and acute graft-vs.-host disease (aGVHD) outcomes. | 100days

SECONDARY OUTCOMES:
Association between donor neutrophil subsets and chronic GVHD (cGVHD) | 6 months
Association between donor neutrophil subsets and leukemia relapse | 6 months
Association between donor neutrophil subsets and non-relapse mortality (NRM) | 6 months
Association between donor neutrophil subsets and disease-free survival (DFS) | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Hua Jin, Principal Investigator — Nanfang Hospital, Southern Medical University
Locations (1):
- Nanfang Hospital, Southern Medical University, Guangzhou, Other (Non U.s.), China

IPD SHARING:
Plan to Share IPD: No